CLINICAL TRIAL: NCT01463722
Title: Study of Accuracy of Amniotic Fluid Lamellar Body Counting for Evaluating of Fetal Lung Maturity
Brief Title: Accuracy of Amniotic Fluid Lamellar Body Counting for Evaluating of Fetal Lung Maturity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, Research Assistant, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASD-1213-20
Record Dates: First submitted 2011-10-30; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Retained Fetal Lung Fluid
Keywords: Respiratory distress syndrome; Lung maturity; lamellar body
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amniotic fluid Lamellar Body Counting (Other)
  Interventions: Other: Amniotic fluid Lamellar Body Counting

INTERVENTIONS:
Other: Amniotic fluid Lamellar Body Counting — fluid samples were obtained by amniocentesis during normal delivery or before rupturing the membrane in cesarean. The samples were sent to the lab as soon as possible and after centrifuging with 500 round per minute for 3 minutes, they were placed in the cell counter machine (STKR coulter).

SUMMARY:
The purpose of this study is to determine the accuracy of Amniotic fluid Lamellar Body Counting for Evaluating of Fetal Lung Maturity.

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) is one of important cause of mortality in neonates. This study was designed to evaluate the amniotic fluid lamellar body counting for predicting fetal lung maturity.

ELIGIBILITY:
Inclusion Criteria:

* Women, with 28-37 weeks of gestational age, who had been decided to terminate their pregnancy, were enrolled in the study

Exclusion Criteria:

* Chorioamnionitis
* Intra Uterine Fetal Death (IUFD)
* Blood in amniotic fluid
* Rupture of placenta and patient dissatisfaction were the exclusion criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The statues of respiratory of neonates | at 2 minutes after delivery
  Diagnosing of immaturity is based on the following criteria: 1-Physical examinations such as: nasal flaring, retraction, grunting, and tachypnea. 2-Oxygen needing more than 24 hours with three chest x-ray findings.

CONTACTS AND LOCATIONS:
Overall Officials: farzaneh memarzadeh, MD, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran